CLINICAL TRIAL: NCT03399747
Title: Phase 2 Study of Abbreviated 3 Cycles of Rituximab Plus CHOP (Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone) Immunochemotherapy in Patients With Completely Excised LocalizedGastrointestinal CD20 (+) Diffuse Large B-cell Lymphoma
Brief Title: Abbreviated 3 Cycles of Rituximab Plus CHOP(Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone) Immunochemotherapy in Patients With Completely Excised LocalizedGastrointestinal CD(Cluster of Differentiation Antigen)20(+) Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Cheolwon Suh, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Asan_LMP2017-002
Record Dates: First submitted 2017-12-25; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abb-R-CHOP (Experimental)
  Interventions: Drug: Abb-R-CHOP

INTERVENTIONS:
Drug: Abb-R-CHOP — Completely Excised LocalizedGastrointestinal CD20 (+) Diffuse Large B-cell Lymphoma
  3 Cycles(1 Cycle:4weeks) of Rituximab Plus CHOP (Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone) Immunochemotherapy

SUMMARY:
Phase 2 Study of Abbreviated 3 Cycles of Rituximab plus CHOP (Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone) Immunochemotherapy in Patients with Completely Excised Localized Gastrointestinal CD20 (+) Diffuse Large B-cell Lymphoma(SATURDAY STUDY)

ELIGIBILITY:
Inclusion Criteria:

* Completely Excised LocalizedGastrointestinal CD20 (+) DLBCL(Diffuse Large B-cell Lymphoma )
* CD 20, CD5, CD10, MUM-1, BCL-6, BCL-2, Ki-76, EBV(Epstein-Barr virus )positive
* Lugano Criteria: Stage I, II1
* Paris Criteria: T1-2NO-1MO
* Stage-adjusted International Prognostic Index: 0-1
* A patient who has not previously received chemotherapy or radiation treatment for the DLBCL
* ECOG(Eastern Cooperative Oncology Group ) :0-2
* In case of patients who do not have any residual lesion due to complete surgical removal of lymphoma I. A patient who has been confirmed to have no residual lesion in the CT conducted following surgery or Ii. Preoperative imaging confirmed as the first phase of a single lesion and post-operative lesion finding that the patient has been confirmed with
* In case of a 50 % or higher cardiac output when there is no clinically significant abnormality in MUGA(multiple gated acquisition scan) or deep frequency
* If appropriate renal function (below serum creatinine 2.0 mg dL or an estimated glomerule filtration rate of 40 mL / mill1.73m2 or higher)
* If the appropriate liver function is present (serum bilirubin), less than three times the normal upper limit of AST(aspartate aminotransferase ) (non-hepatic) unless the serubin is caused by Gilbert syndrome or originated from a non-hepatic ;
* Proper Bone marrow function (ANC-1500mm 3 or higher, number of platelets > 755mm3, and hemoglobin 9.0 g/L or higher) If the screening in the CS(cerebrospinal fluid)F is not acceptable, the dose is given in - 7
* For males, blocking contraceptive methods such as condoms are required at least 6 months from the date of the last administration of the cancer and such measures are agreed
* For fertile women, it must be agreed to apply contraceptive measures (oral contraceptive pills, in the womb, blocking contraceptive methods, etc.) for at least 6 months from the date of administration of the last cancer.
* decided to participate in this study voluntarily and agree in writing

Exclusion Criteria:

* HIV or HCV(hepatitis C virus) positive patient. However, HBVhepatitis B virus) positive patients using anti-viral therapy are allowed
* Patient with current history of other cancers (e.g. cervical carcinoma in situ, treated basal cell carcinoma, early cancer, excluded from the present condition of cancer.
* pregnant or nursing woman, male or female who do not agree with appropriate contraception.
* Systemic disease that is inappropriate for administration of anticancer drugs I. A patient who within the past 6 months had a clinically significant heart attack (non-medical congestive heart failure, symptomatic coronary artery disease, severe myocardial infarction) or Ii. Serious neurology and psychiatric disease Iii. Serious activity infection Iv. Other medical conditions that are difficult to perform in clinical trials
* If you are allergic to chemicals used in this study
* Patients who receive another test medication during a clinical trial or who is administered both chemotherapy, hormone therapy and immunization
* Patient with Bulky disease (length of diaphragm 10 cm)
* Patient who is unsuitable for participation in a clinical examination according to the judgment of a researcher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response | 6 to 8 weeks after completion of the 3rd cycle of treatment(each cycle is 28days)
  CT(Computed tomography) / PET-CT(Positron emission computed tomography)/ Colonoscopy(if necessary) by Lugano stage I or II1, Paris stage T1-2NO-1MO

SECONDARY OUTCOMES:
Assess response rate | after completion of the treatment, up to 2years
  CT/ PET-CT/Colonoscopy(if necessary) by Lugano stage I or II1, Paris stage T1-2NO-1MO
Assess response rate | after completion of the treatment, up to 4years
  CT/ PET-CT/Colonoscopy(if necessary) by Lugano stage I or II1, Paris stage T1-2NO-1MO

OTHER OUTCOMES:
Assess overall survival | after completion of the treatment, up to 5years
  CT/ PET-CT/Colonoscopy(if necessary) by Lugano stage I or II1, Paris stage T1-2NO-1MO